CLINICAL TRIAL: NCT00582010
Title: Effects of Inhaled Nitric Oxide on Ischemia-Reperfusion Injury in Human Liver During Transplantation
Brief Title: Study to Evaluate if Inhaled Nitric Oxide Improves Liver Function After Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mallinckrodt (Industry); University of Washington (Other)
Responsible Party: Principal Investigator, Rakesh Patel, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F070112003
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Reperfusion Injury; Liver Injury
Keywords: ischemia-reperfusion; nitric oxide; inflammation; cell-death; Liver-function post transplantation
MeSH Terms: conditions — Reperfusion Injury; Inflammation | interventions — Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Experimental (Experimental): iNO administration
  Interventions: Drug: inhaled nitric oxide
- 2. Placebo (Placebo Comparator): Placebo (nitrogen)
  Interventions: Drug: nitrogen gas

INTERVENTIONS:
Drug: inhaled nitric oxide — inhaled 80ppm for duration of surgery.
  Other Names: iNO
  Arms: 1. Experimental
Drug: nitrogen gas — inhaled
  Arms: 2. Placebo

SUMMARY:
This blinded, placebo-controlled study will administer inhaled nitric oxide to patients undergoing liver transplantation. The purpose of the study is to test if inhaled nitric oxide prevents liver injury associated with the restoration of blood flow. The premise of the current study is provided by previous studies which document a protective effect of inhaled nitric oxide in this clinical setting.

DETAILED DESCRIPTION:
Specifically, presenting ischemia-reperfusion injury to transplanted livers remains a therapeutic goal in improving liver function and potentially expanding the number of transplantable livers. This study aims to assess the efficacy of inhaled nitric oxide to limit ischemia-reperfusion injury in transplanted livers and by doing so improve liver function post transplantation and decrease patient hospital length of stays.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 19 yr of age scheduled to undergo liver transplantation.

Exclusion Criteria:

* Patients < 19 yr of age
* Patients undergoing re-transplantation or dual organ transplantation
* Patients with underlying pulmonary complications

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh P Patel, PhD, Principal Investigator — University of Alabama at Birmingham; Keith A Jones, MD, Principal Investigator — University of Alabama at Birmingham; Devin E Eckhoff, MD, Principal Investigator — University of Alabama at Birmingham; John S Bynon, MD, Study Director — University of Alabama at Birmingham; Blair Smith, MD, Study Director — University of Alabama at Birmingham; Clark Cross, MD, Study Chair — University of Alabama at Birmingham; Luc Frenette, MD, Study Director — University of Alabama at Birmingham; John D Lang, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Lang JD Jr, Teng X, Chumley P, Crawford JH, Isbell TS, Chacko BK, Liu Y, Jhala N, Crowe DR, Smith AB, Cross RC, Frenette L, Kelley EE, Wilhite DW, Hall CR, Page GP, Fallon MB, Bynon JS, Eckhoff DE, Patel RP. Inhaled NO accelerates restoration of liver function in adults following orthotopic liver transplantation. J Clin Invest. 2007 Sep;117(9):2583-91. doi: 10.1172/JCI31892. PMID 17717604
- [Derived] Lang JD Jr, Smith AB, Brandon A, Bradley KM, Liu Y, Li W, Crowe DR, Jhala NC, Cross RC, Frenette L, Martay K, Vater YL, Vitin AA, Dembo GA, Dubay DA, Bynon JS, Szychowski JM, Reyes JD, Halldorson JB, Rayhill SC, Dick AA, Bakthavatsalam R, Brandenberger J, Broeckel-Elrod JA, Sissons-Ross L, Jordan T, Chen LY, Siriussawakul A, Eckhoff DE, Patel RP. A randomized clinical trial testing the anti-inflammatory effects of preemptive inhaled nitric oxide in human liver transplantation. PLoS One. 2014 Feb 12;9(2):e86053. doi: 10.1371/journal.pone.0086053. eCollection 2014. PMID 24533048

RESULTS

PARTICIPANT FLOW:
Groups:
- 1. Experimental: iNO administration
  inhaled nitric oxide : inhaled 80ppm for duration of surgery.
- 2. Placebo: Placebo (nitrogen)
  nitrogen gas : inhaled
Period: Overall Study
Arm/Group | 1. Experimental | 2. Placebo
Started | 40 | 40
Completed | 40 | 39
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Nitric Oxide; Placebo (Nitrogen Gas): 80 ppm was administered by inhalation for the duration of surgery
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Placebo (Nitrogen Gas) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Full Range); unit: years] | 59 (4) [30 to 72] | 61 [24 to 70] | 60 [24 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 31 | 33 | 64
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Changed Rate of Liver Function Recovery Post-transplantation (Percent Change in AST Levels)
Description: The faster the percent decrease of AST reflect the greater the treatment improved liver function post transplant. A positive percent reflects an decrease; a negative percentage reflects a increase. The rate was calculated by measuring AST levels at baseline and at 96 hours post baseline. (AST levels were lower at 96 hours relative to baseline- positive values in data table indicate percent decrease of AST relative to baseline).
Time Frame: baseline and 96 hours after baseline
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
percentage change from baseline | 83 (14.6) | 86.4 (18)

2. Secondary Outcome: Effect of iNO on Hosptial Length of Stay
Description: number of days subject in hospital after surgery until discharge
Time Frame: from surgery through discharge from hospital
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
days | 9.0 [7.5 to 15.5] | 9.0 [7 to 12.5]

3. Primary Outcome: Changed Rate of Liver Function Recovery Post-transplantation (Percent Change in ALT Levels)
Description: The faster the percent decrease ALT reflect, the greater the treatment improved liver function post transplant. A positive percent reflects an decrease; a negative percentage reflects a increase. . (ALT levels were lower at 96 hours relative to baseline- positive values in data table indicate percent decrease of ALT relative to baseline).
Time Frame: baseline and 96 hours after baseline
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
percentage change from baseline | 62.3 (26.8) | 62.4 (34.9)

4. Primary Outcome: Change in Rate of Liver Function Recovery Post-transplantation (Percent Change in Alkaline Phosphatase Levels)
Description: The faster the percent increase of alkaline phosphatase reflect, the greater the treatment improved liver function post transplant. A positive percent reflects an increase; a negative percentage reflects a decrease.
Time Frame: baseline and 96 hours after baseline
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
percentage change from baseline | 239.7 (672.4) | 55 (96.3)

5. Primary Outcome: Change in Rate of Liver Function Recovery Post-transplantation (Percent Change in Prothrombin Times (PT))
Description: The faster the percent increase of PT reflect, the greater the treatment improved liver function post transplant. A positive percent reflects an decrease; a negative percentage reflects a increase.
Time Frame: baseline and 96 hours after baseline
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
percentage change from baseline | 48.9 (9.9) | 25.5 (37.4)

6. Primary Outcome: Change in Rate of Liver Function Recovery Post-transplantation (Percent Change in Bilirubin Levels)
Description: A positive percent reflects an decrease; a negative percentage reflects a increase.
Time Frame: baseline and 96 hours after baseline
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
percent change from baseline | 6.6 (57) | 0.4 (56.7)

7. Secondary Outcome: Effect of iNO on SICU Stay
Description: Number of minutes after surgery subject remained in SICU
Time Frame: baseline to discharge for SICU
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
minutes | 2533 [1983 to 3075] | 2518 [1703 to 3802]

8. Primary Outcome: Change in Rate of Liver Function Recovery Post-transplantation (Decrease in Hepatobiliary Complications)
Description: Number of complications due to hepatobiliary events.
Time Frame: baseline to 9 months after transplantation
Measure: Number; unit: Complications
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
Complications | 2 | 5

9. Primary Outcome: Number of Complications Related to Liver Function Recovery Post-transplantation (Total Complications) at 9 Months Post Surgery
Description: Number of any complication reported by subjects at 9 months after surgery
Time Frame: baseline to 9 months post surgery
Measure: Number; unit: complications
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 40 | 39
complications | 44 | 83

ADVERSE EVENTS:
Arm/Group | 1. Experimental | 2. Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Experimental (N=40) | 2. Placebo (N=39)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days